CLINICAL TRIAL: NCT06209138
Title: Tailoring of HPMC-Zein Based Film Forming Gel of 5-fluorouracil for Treat-ment of Stable Vitiligo: a Strategy Assisted by Carbon Dioxide Laser Dermabra-sion
Brief Title: 5-fluorouracil for Treatment of Stable Vitiligo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mahmoud A Makki, MD, Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HV04/2020
Record Dates: First submitted 2023-12-22; First posted 2024-01-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Vitiligo
Keywords: 5FU; Film forming gel; vitiligo; JAK3 gene expression; Dermabrasion
MeSH Terms: conditions — Vitiligo | interventions — Fluorouracil; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CO2 laser assisted dermabrasion and 5FU film (Experimental)
  Interventions: Drug: 5 fluorouracil
- CO2 laser assisted dermabrasion and saline (Active Comparator)
  Interventions: Other: Saline

INTERVENTIONS:
Drug: 5 fluorouracil — 5 fluorouracil (5FU) using different ratios of hydroxyl propyl methyl cellulose (HPMC) and Zein
  Arms: CO2 laser assisted dermabrasion and 5FU film
Other: Saline — Normal saline solution contains 0.9 percent sodium chloride (salt)
  Arms: CO2 laser assisted dermabrasion and saline

SUMMARY:
Vitiligo, a significant dermatologic challenge affecting 0.5 to 2% of the global population. Despite various existing medical approaches, current vitiligo treatments are still far from optimal.

DETAILED DESCRIPTION:
Vtiligo, a significant dermatologic challenge affecting 0.5 to 2% of the global population. Despite various existing medical approaches, current vitiligo treatments are still far from optimal. 5FU is a well-known chemotherapeutic agent that has been used for colorectal cancer treatment. The drug prevents DNA synthesis by inhibiting the thymidylate synthetase. The hyperpigmenta-tion of the skin is the most side effect observed with 5-FU therapy which directed its use in treat-ment of vitiligo. Besides, many studies reported that 5-FU could induce regimentation in vitiligo by direct stimulation of melanocytes and increasing melanosomes numbers in the keratinocytes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable vitlligo

Exclusion Criteria:

* patients under the age of 10 years.
* Individuals with a history of the Koebner phenomenon, a tendency for keloid or hypertrophic scarring
* Pregnancy.
* Recent isotretinoin therapy within the last 6 months.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Guartile grading scale | 2 months
  A grading system with a quartile grading scale was used. Here, grading of > 75% will be considered excellent improvement, very good (51-75%), good (50-25%), poor (<25%), mild (25%), and poor improvement if less than 25% grading.
analysis of Jak3 expression in vitiligo lesions | 2months
  the improvement will be associated with a reduction in JAK levels

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Asyut, No State, Egypt

IPD SHARING:
Plan to Share IPD: No